CLINICAL TRIAL: NCT04582643
Title: Validation of a Healthy Metabolic Behavior Tool for Overweight and Obese Women
Brief Title: Pilot Test of a Healthy Metabolic Behaviour Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIRB 2020/2530
Record Dates: First submitted 2020-09-25; First posted 2020-10-09 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Metabolic Disease; Obese; Diet Habit
MeSH Terms: conditions — Metabolic Diseases; Obesity; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Single arm pilot test of lifestyle intervention using newly developed tool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 6P intervention (Experimental): 6P assessment along with education provided based on the 6P components.
  Interventions: Behavioral: 6P intervention

INTERVENTIONS:
Behavioral: 6P intervention — 6P assessment targeting on diet, activity and mentality, along with education provided based on the 6P components. The 6P tool serves the functions to help the women to self-monitor and be aware of their negative lifestyle choices.

SUMMARY:
This study aims to validate and pilot test the short-term intervention effect of a newly developed healthy metabolic behaviour tool, named as the 6P tool, on dietary attitude/ practice and body weight changes over one month among overweight and obese women. A total of 50 women, aged 21-40 years, BMI ≥25 kg/m2, who are attending the preconception clinic and planning for a pregnancy over the next one year, will be invited to participate in this pilot study. The recruitment period is estimated to take up to 10 weeks, with subsequent 1 month follow-up visit.

DETAILED DESCRIPTION:
Preconception is a stage that could critically influence subsequent antenatal and postnatal health of mother and offspring. In Singapore, approximately one-third of women are overweight and obese during the preconception period. In the present pilot study, the investigators aim to introduce a simple, self-administered tool that can identify discrete components of an individual's diet, which would lead to self-awareness, self-evaluation and self-education, and over time, results in a positive change in eating habits and health. Specifically, the study aims i) to validate a newly developed tool that comprises six main dietary components (6P), namely Portion, Proportion, Pleasure, Phase, Physicality and Psychology in overweight and obese women during the preconception period; (ii) and to assess the short-term intervention effect of the 6P tool on dietary attitude/ practice and body weight changes over one month. The investigators hypothesise that intervention using this 6P tool in overweight and obese women will help them to promote healthy eating behaviours and reduce body weight. This study targets to recruit 50 overweight/ obese preconception women, from KK Women's and Children's Hospital, to evaluate the effectiveness of the tool over one month. Throughout the one month follow up period, nudges in the form of text messages/images related to the 6P goals will be sent to participants through mobile phone. This validated 6P tool is planned to be applied in a preconception targeted intervention cohort in order to build a positive mental model in healthy eating among overweight and obese women, enhancing awareness and belief towards weight management behaviour, and promoting a healthy life cycle.

ELIGIBILITY:
Inclusion Criteria:

* age 21-40 years
* body mass index >= 25 kg/m2

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women planning to conceive
Enrollment: 50 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Meal portion size | Between baseline and follow-up visit (1 month)
  Assessed by the portion size rating (scores1-7) in the 6P tool before and after the intervention. Higher score indicates higher portion size.
Vegetable intake | Between baseline and follow-up visit (1 month)
  Assessed by the proportion assessment for vegetable intake in the 6P tool before and after the intervention
Pleasure food intake | Between baseline and follow-up visit (1 month)
  Assessed by the frequency of pleasure food intake in the 6P tool before and after the intervention
Meal timing | Between baseline and follow-up visit (1 month)
  Assessed by the percentage of total caloric intake during the day and night in the 6P tool before and after the intervention
Physical activity | Between baseline and follow-up visit (1 month)
  Assessed by the duration of physical activity in the 6P tool before and after the intervention
Motivational level | Between baseline and follow-up visit (1 month)
  Assessed by the rating of motivational level (scores 1-9) in the 6P tool before and after the intervention. Higher score indicates higher motivational level.

SECONDARY OUTCOMES:
Body weight changes | Between baseline and follow-up visit (1 month)
  Weight changes in kg before and after the intervention
Body mass index changes | Between baseline and follow-up visit (1 month)
  Body mass index changes in kg/m2 before and after the intervention
Dietary behavioral changes | Between baseline and follow-up visit (1 month)
  Assessed by the Three Factor Eating Questionnaire before and after the intervention
Activity intensity changes | Between baseline and follow-up visit (1 month)
  Assessed by the International Physical activity Questionnaire
Screen viewing time changes | Between baseline and follow-up visit (1 month)
  Assessed by the Sedentary Behavioural Questionnaire

OTHER OUTCOMES:
Clarify, usefulness and acceptability of the 6P tool | Follow up visit at 1 month
  Assessed by the feedback evaluation questionnaire
Usefulness and acceptability for the nudges | 1 month
  Assessed by the nudges rating scale and feedback evaluation questionnaire
Other lifestyle changes | Between baseline and follow-up visit (1 month)
  Assessed by the general lifestyle questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Kok Yen Chan, PhD, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No